CLINICAL TRIAL: NCT04064164
Title: SPEEKO for Elderspeak: A Self-Monitoring App to Improve Communication and Reduce Behavioral Symptoms in Care for Persons With Alzheimer's Disease and Other Dementias
Brief Title: Speeko for Elderspeak: A Self-Monitoring App to Improve Nursing Home Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R21AG065029 (NIH); R21AG065029 (NIH)
Record Dates: First submitted 2019-08-16; First posted 2019-08-21 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Dementia; Staff Attitude
Keywords: Nursing home; Dementia; Technology
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Six nursing homes will be randomly assigned to treatment and control conditions. All NHs will received the CHATO training. The treatment NHs will received immediate feedback from the Speeko App after each recording sessions whereas the Control NHs will not receive feedback until all recording sessions are complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The treatment NHs will received immediate feedback from the Speeko App after each recording sessions
  Interventions: Behavioral: Speeko for Elderspeak
- Control (No Intervention): The Control NHs will not receive app feedback until all recording sessions are complete.

INTERVENTIONS:
Behavioral: Speeko for Elderspeak — Speeko for Elderspeak is a communication feedback IOS application.
  Arms: Treatment

SUMMARY:
This study will test feasibility and preliminary effects of an automated and performance-based feedback app (Speeko for Elderspeak) that detects and reports the use of diminutives (terms of endearment such as honey, dearie, and sweetie), prevalent elderspeak terms linked to BPSD. Building on proof of concept established in the laboratory, the app will demonstrate feasibility at the point-of-care. Next, a clinical trial (N= 6NHs) will be conducted to test preliminary efficacy of the app for amplifying reductions in diminutives use for NH staff completing the CHATO training (3 online modules).

DETAILED DESCRIPTION:
A new person is diagnosed with Alzheimer's disease or other dementia every 66 seconds, and most persons with dementia (PWD) spend the late stages of dementia in nursing homes (NHs) where lack of dementia care skills and staff shortages limit quality of care. Care of PWD in NHs is complicated by behavioral and psychological symptoms of dementia (BPSD) such as aggression, vocal outbursts, wandering, and withdrawal that occur as PWD lose cognitive and communication abilities and cannot express their unmet physical and psychosocial needs. BPSD present to NH staff as resistiveness to care (RTC) that increases staff stress and costly time to complete care, often leading to staff turnover, injury, and inappropriate use of psychotropic medications to control BPSD. Although Center for Medicare and Medicaid Services (CMS) mandates and penalties have reduced antipsychotic medication use slightly, contraindicated use in NH residents remains a pervasive problem, causing harmful side effects and reducing the quality of life for PWD.

The PI and other researchers have empirically verified that RTC occurs when NH staff use elderspeak (speech similar to baby talk) that features inappropriately intimate terms of endearment (diminutives such as "honey"), belittling pronoun substitutions that imply dependence ("the investigators" need a bath), and harsh task-oriented commands ("sit down"). Elderspeak conveys a message of disrespect and incompetence to residents who react with withdrawal or BPSD. The R03 study established that residents with dementia are more than twice as likely to exhibit BPSD (measured by coding RTC behavior in videos) when staff use elderspeak instead of normal adult communication. The subsequent CHAT R01 trial verified that staff reduced their use of elderspeak after attending the three-session Changing Talk (CHAT) communication training program, and that this reduced RTC.

To facilitate dissemination, interactive online CHAT modules have been developed (CHATO) which provides the same CHAT classroom content with the advantage of flexible access via the internet for busy NH staff, including those in rural areas and small, independent NHs. Recognizing the delay and incomplete adoption and application of evidence-based skills in practice, the PI and colleagues believe additional strategies to optimize CHATO skills implementation are indicated. Performance-based reinforcement of skills is effective in achieving greater immediate implementation and long-term maintenance of new skills use in practice. However, feasibility and costs for individualized expert feedback in NH settings are usually prohibitive and thus not widely used in practice.

This study will test feasibility and preliminary effects of an automated and performance-based feedback app that detects and reports the use of diminutives (terms of endearment such as honey, dearie, and sweetie) which are prevalent elderspeak terms linked to BPSD. The PI and colleagues developed the SPEEKO for Elderspeak app using archived NH recordings from previous research to identify the most commonly used diminutives and then to develop algorithms to detect them in speech. Building on proof of concept established in the laboratory, the app will demonstrate feasibility at the point-of-care. Next, a clinical trial (N= 6NHs) will be conducted to test preliminary efficacy of the app for amplifying reductions in diminutives use for NH staff completing the CHATO training.

SPECIFIC AIMS:

1. AIM 1. Demonstrate feasibility, acceptability, and validity of the SPEEKO for Elderspeak feedback app use by staff in the NH. Five certified nursing assistants (CNAs) will use the app during NH care and provide feedback about any needed modifications. Hypothesis: The app will be readily used and acceptable to CNAs. Diminutive counts determined by the app will be correlated with psycholinguistic analysis, validating accuracy.
2. AIM 2. Test preliminary effects of an innovative self-monitoring feedback app on staff elderspeak use and compare accuracy to psycholinguistic analyses of audio-recorded staff communication. Hypothesis: Staff who receive immediate app feedback (N= 30 in three NHs) will have greater elderspeak reduction after completing CHATO training compared to delayed feedback controls (N= 30 in three NHs).
3. AIM 3. Evaluate app acceptability and costs. Hypothesis: Staff who use the app will find it acceptable and beneficial for their practice. Process-based costing will be used to determine costs for app use in NHs and other long-term service and support settings. Costs will be compared in relation to each group's outcomes.

ELIGIBILITY:
Inclusion Criteria:

* CNAs who are age 18 or older
* Permanent employees
* Fluent in English

Exclusion Criteria:

* CNAs younger than 18 or
* CNAs who are not fluent in English.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Williams, RN, PhD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas School of Nursing, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Share study information vis Open Science Framework, platform created by Center for Open Science
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be shared within one year of study completion.
Access Criteria: https://cos.io/our-products/osf/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to the COVID-19 Pandemic, only one nursing home participated. Individual staff members were assigned to groups, however, most withdrew due to extreme turnover.
Groups:
- Treatment: The NH staff participants will received immediate feedback from the Speeko App after each recording sessions
  Speeko for Elderspeak: Speeko for Elderspeak is a communication feedback IOS application.
- Control: The NH staff participants will not receive app feedback until all recording sessions are complete.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 10 | 10
Completed | 2 | 2
Not Completed | 8 | 8
Not completed — Withdrawal by Subject | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 0 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Elderspeak Measured by Diminutives Detected in Participant's Recorded Speech.
Description: Diminutive Use per Utterance detected by the Speeko for Elderspeak app. Diminutive data will be compared between the intervention and control groups and within nursing homes. The clinical trial could not be analyzed due to too few participants (COVID-19 Pandemic).
Time Frame: Time1(baseline), Time 2 (immediately post-1 week CHATO training), Time 3 (2 weeks post-CHATO), Time 4 (4 weeks post-CHATO)
Measure: Mean (Standard Deviation); unit: Diminutive Use per Utterance
Arm/Group | Treatment | Control
Number analyzed (Participants) | 2 | 2
Diminutive Use per Utterance
  Time 1 | 0.03 (0.01) | 0.00 (0.01)
  Time 2 | 0.00 (0.00) | 0.01 (0.01)
  Time 3 | 0.01 (0.00) | 0.00 (0.00)
  Time 4 | 0.01 (0.01) | 0.01 (0.01)

2. Secondary Outcome: Acceptability as Measured by System Usability Scale.
Description: A validated, 10-item industry standard survey. Questions are in 5-point Likert scale with responses from strongly agree to strongly disagree. Question scores are converted to a 0-100 total score where lower scores indicate low usability and high scores indicate greater usability. A single value was calculated by summing all scores across and averaged.
Time Frame: Survey completed after using the Speeko app during a feasibility session (pre-clinical trial) or at the end of all four recording sessions - Time 4 (4 weeks post-CHATO).
Measure: Mean (Standard Deviation); unit: units on a scale 0-100
Groups:
- Survey Participants: Seven participants rated the SPEEKO for Elderspeak app using the System Usability Scale.
Arm/Group | Survey Participants
Number analyzed (Participants) | 7
units on a scale 0-100 | 69.9 (14.6)

3. Secondary Outcome: Evaluate the App Cost by Measuring Wages Per Hour by NH Role and Costs Associated With the Speeko for Elderspeak Application.
Description: The cost associated with elderspeak reduction will be calculated using primary outcomes, wage data, and application costs.
Time Frame: The survey was completed by each nursing home at the end of the 3-month implementation period.
Population: Due to the COVID-19 pandemic only 4 people completed the clinical trial. The data were not collected.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

4. Post Hoc Outcome: The Number of Elderspeak Diminutives Detected in Participant's Recorded Speech.
Description: The number of diminutives detected by the Speeko for Elderspeak app will be correlated with manual psycholinguistic analysis to determine app accuracy. Diminutive data will be compared between the intervention and control groups and within nursing homes.
Time Frame: Only the baseline data was analyzed for all participants enrolled in the study.
Population: The baseline data was analyzed for 25 participants. Recordings for the participants were analyzed to compare elderspeak detected by human vs. computer (Speeko App) detection.
Measure: Number; unit: Number of Diminutive Words Identified
Groups:
- Baseline Data for All Groups Plus Feasibility - Human Identification: Testing was completed during 2020 for the first NH (n= 5) and during 2022 for the second NH (n=20). Testing was interrupted by the COVID-19 pandemic and restricted access and severe staffing shortages and use of temporary staff during and at the end of the pandemic.
  Diminutives were identified by human coders
- Baseline Data for All Groups Plus Feasibility - App Identification: Testing was completed during 2020 for the first NH (n= 5) and during 2022 for the second NH (n=20). Testing was interrupted by the COVID-19 pandemic and restricted access and severe staffing shortages and use of temporary staff during and at the end of the pandemic.
  Diminutives were identified by the Speeko for Elderspeak App.
Arm/Group | Baseline Data for All Groups Plus Feasibility - Human Identification | Baseline Data for All Groups Plus Feasibility - App Identification
Number analyzed (Participants) | 25 | 25
Number of Diminutive Words Identified
  Dear | 36 | 18
  Sweet | 23 | 10
  Girl | 47 | 22
  Honey | 49 | 38
  Baby | 15 | 15
Statistical Analysis 1: Comparison: Baseline Data for All Groups Plus Feasibility - Human Identification vs Baseline Data for All Groups Plus Feasibility - App Identification; Test type: Equivalence — Pearson's Chi-square test was completed between the total instances of diminutives either identified by human or the Elderspeak App; p = .004, Chi-squared — Dear (root word); X-squared = 8.4 df=1
Statistical Analysis 2: Comparison: Baseline Data for All Groups Plus Feasibility - Human Identification vs Baseline Data for All Groups Plus Feasibility - App Identification; Test type: Equivalence — Pearson's Chi-square test was completed between the total instances of diminutives either identified by human or the Elderspeak App. Significant associations indicated the human and app were accurately identifying true positives (1:1) or true negatives (0:0); p < .001, Chi-squared — Sweet (root word); X-squared = 20.20 df=1
Statistical Analysis 3: Comparison: Baseline Data for All Groups Plus Feasibility - Human Identification vs Baseline Data for All Groups Plus Feasibility - App Identification; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = .02, Chi-squared — Girl (root word); X-squared = 5.08, df=1
Statistical Analysis 4: Comparison: Baseline Data for All Groups Plus Feasibility - Human Identification vs Baseline Data for All Groups Plus Feasibility - App Identification; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = .10, Chi-squared — Honey (root word); X-squared = 2.7, df= 1
Statistical Analysis 5: Comparison: Baseline Data for All Groups Plus Feasibility - Human Identification vs Baseline Data for All Groups Plus Feasibility - App Identification; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.85, Chi-squared — Baby (root word); X-squared = 12.2, df = 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT04064164/Prot_SAP_000.pdf